CLINICAL TRIAL: NCT06054516
Title: Hyperpolarized MRSI in Ischemic Heart Disease: Metabolic Profiling of the Myocardium
Brief Title: Hyperpolarized MRSI in Ischemic Heart Disease: A Metabolic Investigation of the Heart Muscle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henrik Wiggers (Other)
Responsible Party: Sponsor-Investigator, Henrik Wiggers, Professor, PhD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: 65424
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ischemic heart disease
  Interventions: Diagnostic Test: 13C-enriched pyruvate

INTERVENTIONS:
Diagnostic Test: 13C-enriched pyruvate — Before starting the hyperpolarization injection procedure, the patient will be scanned using the standard MR imaging defined in the clinical protocol and 13C prescriptions and a pre-scan will be completed. The clinical investigator will mount the administration syringe in the MR compatible power-injector with pre-adjusted injection volume calculated according to body weight (0.43 ml /kg bw). This setting is checked by the scanning operator and clinical investigator. The injection valve is set for agent delivery, and agent injected at a rate of 5 ml/s. The timings are monitored using a stopwatch on the SPINLAB. Following injection of hyperpolarized [1-13C]-Pyruvate , 20 ml of sterile saline in a separate syringe, already attached to the patient line, will be used to flush the IV line at the same injection rate (5 ml/s).

SUMMARY:
This study aims to investigate the potential of using hyperpolarized [1-13C]-pyruvate magnetic resonance imaging (MRI) to assess metabolic alterations in patients with ischemic heart disease (IHD). Altered myocardial metabolism is recognized as a crucial factor in heart failure and IHD, and modulating cardiac metabolism offers a new approach to treatment. However, current diagnostic modalities use ionizing radiation and have shown limited prognostic value.

Hyperpolarization through dynamic nuclear polarization (DNP) enables highly sensitive in vivo detection of metabolic processes. Hyperpolarized [1-13C]-pyruvate allows visualization of glycolysis-related metabolism, providing insights into the breakdown of glucose and its derivatives. By using this technique, the study aims to differentiate viable from non-viable myocardium in patients with IHD.

The objectives include implementing hyperpolarized [1-13C]-pyruvate cardiac MRI to image metabolic flux in the human heart and investigating the potential of this method to distinguish viable from non-viable myocardium in patients with IHD. The study endpoints involve assessing metabolic flux through the pyruvate dehydrogenase complex (PDC) and analyzing ratios of different metabolites, which can indicate the extent of pyruvate oxidation and lactate production.

A cross-sectional study design involving patients with CHF and ischemic heart disease will be used. Patients will undergo hyperpolarized [1-13C]-pyruvate MRI, PET imaging, late gadolinium enhancement (LGE) MRI, and cardiac magnetic resonance imaging (CMR). The study will compare [1-13C]-pyruvate MRI findings with PET results, allowing for a correlation between metabolic data and traditional imaging techniques. This innovative approach could provide valuable insights into the metabolic changes associated with ischemic heart disease

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure
* >18 years of age
* Left ventricular Ejection Fraction (LVEF) of 10 - 60 %
* Adequate hematologic and organ function.
* Women who are not postmenopausal or surgically sterile must have a negative serum or urine pregnancy test performed at time of inclusion in the study.
* Safe and highly effective contraception must be used throughout the study meaning either hormonal anti-conception or an anti-fertility intrauterine device. If the partner is non fertile or the patient has no sexual activities, this is also accepted.
* Non-insulin dependent Diabetes mellitus is allowed
* Danish speaking
* Able and willing to comply after informed consent
* Ischemic heart disease and referral to viability testing at the Department of Clinical Physiology and Nuclear Medicine at Aarhus University Hospital.

Exclusion Criteria:

* Not able or willing to receive heart failure therapy
* Patients not willing to participate
* Uncontrolled serious medical condition, such as uncontrolled heart disease, uncontrolled diabetes, intestinal obstruction, uncontrolled hypertension, or recent cerebral ischemia
* Estimated Glomerular Filtration Rate (eGFR) <30 mL/min
* Insulin dependent Diabetes Mellitus
* Intolerance to Pyruvate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease treated at Aarhus University Hospital
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative numerical data given as metabolite ratios | 45 minutes
  [13C]-bicarbonate/[1-13C]-pyruvate ratio, b) [1-13C]-lactate / [1-13C]-pyruvate ratio and [1-13C]-lactate / [1-13C]-bicarbonate ratio. The latter gives ratio indices of PDC-mediated pyruvate oxidation and lactate production via lactate dehydrogenase.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neubauer S. The failing heart--an engine out of fuel. N Engl J Med. 2007 Mar 15;356(11):1140-51. doi: 10.1056/NEJMra063052. No abstract available. PMID 17360992
- [Background] Rider OJ, Tyler DJ. Clinical implications of cardiac hyperpolarized magnetic resonance imaging. J Cardiovasc Magn Reson. 2013 Oct 8;15(1):93. doi: 10.1186/1532-429X-15-93. PMID 24103786
- [Background] Ardenkjaer-Larsen JH, Fridlund B, Gram A, Hansson G, Hansson L, Lerche MH, Servin R, Thaning M, Golman K. Increase in signal-to-noise ratio of > 10,000 times in liquid-state NMR. Proc Natl Acad Sci U S A. 2003 Sep 2;100(18):10158-63. doi: 10.1073/pnas.1733835100. Epub 2003 Aug 20. PMID 12930897
- [Background] Golman K, Petersson JS, Magnusson P, Johansson E, Akeson P, Chai CM, Hansson G, Mansson S. Cardiac metabolism measured noninvasively by hyperpolarized 13C MRI. Magn Reson Med. 2008 May;59(5):1005-13. doi: 10.1002/mrm.21460. PMID 18429038
- [Background] Schroeder MA, Lau AZ, Chen AP, Gu Y, Nagendran J, Barry J, Hu X, Dyck JR, Tyler DJ, Clarke K, Connelly KA, Wright GA, Cunningham CH. Hyperpolarized (13)C magnetic resonance reveals early- and late-onset changes to in vivo pyruvate metabolism in the failing heart. Eur J Heart Fail. 2013 Feb;15(2):130-40. doi: 10.1093/eurjhf/hfs192. Epub 2012 Dec 19. PMID 23258802
- [Background] Cunningham CH, Lau JY, Chen AP, Geraghty BJ, Perks WJ, Roifman I, Wright GA, Connelly KA. Hyperpolarized 13C Metabolic MRI of the Human Heart: Initial Experience. Circ Res. 2016 Nov 11;119(11):1177-1182. doi: 10.1161/CIRCRESAHA.116.309769. Epub 2016 Sep 15. PMID 27635086
- [Background] Hansen ESS, Tougaard RS, Norlinger TS, Mikkelsen E, Nielsen PM, Bertelsen LB, Botker HE, Jorgensen HS, Laustsen C. Imaging porcine cardiac substrate selection modulations by glucose, insulin and potassium intervention: A hyperpolarized [1-13 C]pyruvate study. NMR Biomed. 2017 Jun;30(6). doi: 10.1002/nbm.3702. Epub 2017 Feb 10. PMID 28186677
- [Background] Apps A, Lau JYC, Miller JJJJ, Tyler A, Young LAJ, Lewis AJM, Barnes G, Trumper C, Neubauer S, Rider OJ, Tyler DJ. Proof-of-Principle Demonstration of Direct Metabolic Imaging Following Myocardial Infarction Using Hyperpolarized 13C CMR. JACC Cardiovasc Imaging. 2021 Jun;14(6):1285-1288. doi: 10.1016/j.jcmg.2020.12.023. Epub 2021 Feb 10. No abstract available. PMID 33582059